CLINICAL TRIAL: NCT00499889
Title: Imatinib Mesylate, Busulfan, Fludarabine, Antithymocyte Globulin and Allogeneic Stem Cell Transplantation for Chronic Myelogenous Leukemia
Brief Title: Imatinib Mesylate, Busulfan, Fludarabine, and Antithymocyte Globulin for CML Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Support issue.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID02-901
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Leukemia
Keywords: Chronic Myelogenous Leukemia; Allogeneic Stem Cell Transplantation; Leukemia; Imatinib Mesylate; Gleevec; Busulfan; Busulfex; Myleran; Fludarabine; ATG; STI571; Antithymocyte Globulin; Thymoglobulin
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; fludarabine; fludarabine phosphate; Busulfan; Antilymphocyte Serum; thymoglobulin; Tacrolimus; Methotrexate; Blood Component Removal; Stem Cell Transplantation; Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib, Busulfan, Fludara + Antithymocyte Globulin (Experimental): Oral Imatinib Mesylate 400 mg twice a day for 9 Days; Busulfan 130 mg/m^2 by vein (IV) daily for 2 Days; Fludara 40 mg/m^2 IV daily for 4 Days; Antithymocyte Globulin (ATG) 2.5 mg/kg IV daily for 3 Days; Tacrolimus levels maintained between 5-15 ng/dl, Day -2 to Day 180; Methotrexate 5 mg/m2 on days 1, 3, 6 and 11; and Donor bone marrow or blood stem cells infused on day 0 with possible donor lymphocyte infusion (DLI) for progressive disease.
  Interventions: Drug: Imatinib Mesylate; Drug: Fludarabine (Fludara); Drug: Busulfan; Drug: Antithymocyte Globulin (ATG); Drug: Tacrolimus; Drug: Methotrexate; Procedure: Donor lymphocyte infusion (DLI); Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Imatinib Mesylate — 400 mg by mouth twice daily for 9 Days
  Other Names: Gleevec; STI571
Drug: Fludarabine (Fludara) — 40 mg/m^2 by vein daily for 4 Days
  Other Names: Fludarabine Phosphate; Fludara; Fludarabine
Drug: Busulfan — 130 mg/m^2 by vein daily for 2 Days
  Other Names: Busulfex; Myleran
Drug: Antithymocyte Globulin (ATG) — 2.5 mg/kg by vein daily for 3 Days
  Other Names: ATG; Thymoglobulin
Drug: Tacrolimus — Tacrolimus levels maintained between 5-15 ng/dl, first as continuous IV infusion, and converted to oral every 12 hour dosing as tolerated. Starting day -2 until day 180.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 on days 1, 3, 6 and 11.
Procedure: Donor lymphocyte infusion (DLI) — Infusion of lymphocytes from the original bone marrow donor by vein if relapse after >4 weeks of imatinib.
  Other Names: buffy coat fusion; donor leukocyte infusion; apheresis; donor immune cell infusion
Procedure: Stem Cell Transplant — Infusion of donor bone marrow or blood stem cells by vein over approximately one hour on day 0.
  Other Names: stem cell infusion; stem cell transplantation; ALLOGENEIC STEM CELL TRANSPLANTATION; HSCT; hematopoietic stem cell transplant; Bone Marrow transplant; PBSC; Peripheral Blood Stem Cell

SUMMARY:
Primary Objective:

To estimate the probability of molecular complete remission at one year for the described sequential treatment approach, with nonablative hematopoietic transplantation, post transplant imatinib mesylate and donor lymphocyte infusion, in patients with Ph-positive Chronic Myelogenous Leukemia (CML) not in blastic transformation.

Secondary Objective:

Response to post transplant Imatinib mesylate therapy for 12 weeks as treatment of residual disease, response to donor lymphocyte infusion (DLI) for residual disease following imatinib mesylate therapy, as well as engraftment, toxicity, disease free survival and survival, effect of busulfan pharmacokinetics on study outcome.

DETAILED DESCRIPTION:
Patients will have blood and bone marrow tests performed as well as chest and sinus X-rays and tests of their heart and lung function. Approximately 5 tablespoons of blood will be drawn.

All patients in this study will receive imatinib mesylate by mouth for 9 days, unless the patient is known to be allergic or have symptomatic intolerance to the drug, or if the leukemia has failed to respond to imatinib. Fludarabine 40 mg/m2 by vein for 4 days (days -5 to -2), busulfan 130 mg/m2 by vein for 2 days (days -3 and -2), and ATG (Antithymocyte Globulin) 2.5 mg/kg by vein for 3 days (-3,-2 and -1).

Patients will then receive the donor bone marrow or blood stem cells by vein over approximately one hour on day 0.

After the infusion of the donor cells, you will receive immunosuppressive therapy with tacrolimus and methotrexate to decrease the risk of developing graft-vs-host disease (GvHD).

Patients will need frequent blood tests to monitor their counts and blood chemistries. This is generally done daily while in hospital and at least twice per week for the first 100 days post transplant. You may need frequent blood transfusions and may have to be admitted to the hospital to receive antibiotics if they develop fever. Bone marrow will be examined frequently beginning four weeks after treatment to evaluate response to treatment; Blood and bone marrow exams are to be performed at one, two three, six, 12 and 18 months post transplant and yearly thereafter for 5 years. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle.

Patients in whom treatment produces a remission, in which no sign of the leukemia can be detected, will receive no further therapy unless the leukemia recurs. Patients with evidence of leukemia after 3 months from the transplant will receive additional treatment with imatinib mesylate; those with detectable leukemia after an additional 3 months may receive an infusion of immune cells from the transplant donor.

If there is evidence of leukemia after the transplant, you will receive additional treatment with imatinib mesylate. If leukemia cells can still be detected, additional donor immune cells will be given to you by vein.

Patients are considered on the study for 5 years after the transplant.

A total of 90 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Ph+ chronic myelogenous leukemia (CML) in first chronic phase without a complete hematologic response after 3 months of Imatinib mesylate therapy, or >=35% Ph+ cells despite > 6 months of Imatinib mesylate treatment, or after disease progression from a complete or partial response. Any patient with accelerated phase or blast crisis who achieves a subsequent chronic phase is eligible. Patients must have an HLA matched related or unrelated donor or one antigen mismatched related donor.
2. Patients should be less than 70 years of age. Patients less than 30 years of age who achieve a hematologic remission with imatinib therapy are eligible regardless of cytogenetic response.
3. Patients are stratified as Group 1: First chronic phase, Group 2 Accelerated phase or blast crisis that achieved a hematologic remission with imatinib mesylate-based treatment.

Exclusion Criteria:

1. Zubrod Performance Scale (PS) >=2, uncontrolled infection, Creatinine > 2.0 mg/dl; Ejection fraction < 40%; Carbon Monoxide Diffusing Capacity (DLCO) < 45% of predicted; Serum bilirubin > 2 gm/dl; GPT (Glutamic-pyruvic transaminase) or GOT (glutamic-oxaloacetic transaminase)> 3 times normal values. Patients should not be human immunodeficiency virus (HIV) seropositive or pregnant.
2. Patients should not have progressed to accelerated phase or blast crisis while receiving imatinib mesylate containing therapy.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 02/12/03 to 01/15/09. All patients were recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: One patient registered for transplant became ineligible before any treatment due to infection and was taken off study; 41 patients received the transplant regimen and an Allogeneic transplant.
Groups:
- Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin: Oral Imatinib Mesylate 400 mg twice a day for 9 Days; Busulfan 130 mg/m^2 by vein (IV) daily for 2 Days; Fludara 40 mg/m^2 IV daily for 4 Days; Antithymocyte Globulin (ATG) 2.5 mg/kg IV daily for 3 Days; Tacrolimus levels maintained between 5-15 ng/dl, Day -2 to Day 180; Methotrexate 5 mg/m2 on days 1, 3, 6 and 11; and Donor bone marrow or blood stem cells infused on day 0 with possible donor lymphocyte infusion (DLI) for progressive disease.
Period: Overall Study
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Started | 42
Completed | 41
Not Completed | 1
Not completed — Infection prior to treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 39
  >=65 years | 2
Age Continuous [Median (Full Range); unit: years] | 42.2 (42) [14 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Secondary Outcome: Participants' With mCR Response to Post Transplant Imatinib Mesylate Therapy
Description: Number of participants with response of molecular complete remission (mCR) to Imatinib Mesylate therapy as treatment for residual disease after transplant. Molecular remission is a complete remission with no evidence of disease in the blood cells and/or bone marrow using sensitive polymerase chain reaction (PCR) tests.
Time Frame: 1 Year
Population: Analysis was per protocol. Only 19 participants having the post transplant Imatinib Mesylate Therapy out of the 41 participants treated were analyzed for this outcome.
Measure: Number; unit: Participants
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Number analyzed (Participants) | 19
Participants | 10

2. Primary Outcome: Number of Participants in Complete Molecular Remission at 1 Year
Description: Participants at 1 year in molecular remission, post transplant, post imatinib mesylate and donor lymphocyte infusion (DLI). Molecular remission is a complete remission with no evidence of disease in the blood cells and/or bone marrow using sensitive polymerase chain reaction (PCR) tests (this test is most commonly used in clinical trials).
Time Frame: Baseline to 1 year
Population: Analysis was per protocol. One patient did not receive treatment and was excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Number analyzed (Participants) | 41
participants | 21

3. Secondary Outcome: Participants' With mCR Response to Post Transplant DLI
Description: Number of participants with response of molecular complete remission (mCR) to DLI as treatment for residual disease after transplant. Molecular remission is a complete remission with no evidence of disease in the blood cells and/or bone marrow using sensitive polymerase chain reaction (PCR) tests.
Time Frame: 1 year
Population: Only 8 participants having the post-transplant DLI out of the 41 participants treated were analyzed for this outcome.
Measure: Number; unit: Participants
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Number analyzed (Participants) | 8
Participants | 4

ADVERSE EVENTS:
Time Frame: 5 years and 6 months
Arm/Group | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin
Serious Adverse Events (participants affected / at risk) | 12/41
Other Adverse Events (participants affected / at risk) | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin (N=41)
severe anemia (Blood and lymphatic system disorders) | 1 (1)
increased bilirubin (Hepatobiliary disorders) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2)
neurologic (Nervous system disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Distention (Gastrointestinal disorders) | 1 (1)
Hypertensive Crisis (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Myelosupression (Blood and lymphatic system disorders) | 1 (1)
GVHD (Immune system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesylate, Busulfan, Fludarabine + Antithymocyte Globulin (N=41)
Granulocytes (Blood and lymphatic system disorders) | 1 (1)
platelets (Blood and lymphatic system disorders) | 1 (1)
increased blood pressure (Cardiac disorders) | 1 (1)
increased prothrombin time (Blood and lymphatic system disorders) | 1 (1)
fever (Infections and infestations) | 4 (4)
fatigue (General disorders) | 1 (1)
Gastrointestional Disorder (other) (Gastrointestinal disorders) | 2 (2)
esophagitis (Gastrointestinal disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 4 (4)
diarrhea (Gastrointestinal disorders) | 1 (1)
increased alanine aminotransferase (ALT) (Hepatobiliary disorders) | 1 (1)
increased LDH (Hepatobiliary disorders) | 1 (1) — Lactate dehydrogenase (LDH or LD)
infection (Infections and infestations) | 6 (6)
decreased neutrpoenia (Infections and infestations) | 1 (1)
neurolgic other (Nervous system disorders) | 2 (2)
headache (Nervous system disorders) | 1 (1)
drowiness (Nervous system disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
skin other (Skin and subcutaneous tissue disorders) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Study completed early due to support issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No